CLINICAL TRIAL: NCT03201354
Title: Efficacy and Safety of the ExPRESS Implant Versus Deep Sclerectomy in Combined Surgery: Prospective, Multi-center, Comparative Study
Brief Title: Efficacy and Safety of the ExPRESS Implant Versus Deep Sclerectomy in Combined Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Catala de Retina (Other)
Collaborators: Gregorio Marañón Hospital (Other); Clinica Universidad de Navarra, Universidad de Navarra (Other); Hospital Vall d'Hebron (Other); Hospital Universitario Ramon y Cajal (Other); Hospital San Eloy (Unknown); Hospital del Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICR-01 Ex-PRESS
Record Dates: First submitted 2011-12-21; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Ocular hypertension; Filtration surgery; Trabeculectomy with Ex-PRESS; Non penetrating deep sclerectomy; Phacoemulsification; Combined surgery
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Filtering Surgery; Cataract Extraction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Filtration surgery with Express (Active Comparator): Filtration surgery with Ex-PRESS + cataract extraction (Cataract surgery and IOL implantation)
  Interventions: Procedure: Filtration surgery with Ex-PRESS; Procedure: Cataract extraction
- Non penetrating surgery (Active Comparator): - Filtration surgery with Non penetrating deep sclerectomy + cataract extraction (Cataract surgery and IOL implantation)
  Interventions: Procedure: Non penetrating deep sclerectomy; Procedure: Cataract extraction

INTERVENTIONS:
Procedure: Filtration surgery with Ex-PRESS — Filtration surgery with Ex-PRESS
  Arms: Filtration surgery with Express
Procedure: Non penetrating deep sclerectomy — Non penetrating deep sclerectomy
  Arms: Non penetrating surgery
Procedure: Cataract extraction — Cataract surgery and IOL implantation

SUMMARY:
The Ex-PRESS Glaucoma Filtration Device is a small, non-valved implant that was designed to lower intraocular pressure (IOP) by shunting aqueous humor from the anterior chamber into the subconjunctival space. The implant was developed in response to the need for more straightforward, standardized and safe surgical technique than standard filtration surgery. No iridectomy and no sclerectomy is needed if an Ex-PRESS device is implanted under a partial-thickness scleral flap. This may reduce surgical time and complications when compared to a standard trabeculectomy.

In some studies it has been found to be safe and effective with few complications, even in high-risk patients. No previous studies have compared filtration surgery with Ex-Press implant to deep sclerectomy.

DETAILED DESCRIPTION:
Hypothesis:

In combined procedure (cataract and filtering surgery), the effect of Ex-PRESS device has similar efficacy reducing intraocular pressure than non penetrant deep sclerectomy and with good level of safety.

Objective:

To evaluate and compare the efficacy and safety at 12 months of the filtering surgery with the Ex-PRESS device with that of deep sclerectomy.

Methods:

Design: Multi-center, prospective, simple-blind, randomized study.

Primary variable:

1. Intraocular pressure.

Secondary variables:

1. Success rate at IOP <18
2. Frequency and type of complications
3. Number of hypotensive drugs needed.

Sample size calculation: Accepting an alfa risk of 0.05 and a beta risk of 0.20 in a two-sided Student's T-test, 50 subjects are necessary in first group and 50 in the second to recognize as statistically significant a difference greater than or equal to 10% in IOP, with a common standard deviation of 17%. A drop-out rate of 8% has been anticipated. If no drop-out rate is considered, the number of needed subjects is 92 (46 per group).

If the drop out rate is more than 8%:

1. If the recruitment period is open, another subjects will be included.
2. If the recruitment period os close, the inclusion of another subject will be evaluated to maintain the statistic power of the study.

Method

-Single blinded. Each patient will be assigned to one of the two arms (Ex-PRESS or Deep sclerectomy) the same day of surgery. The surgeon will be informed of the randomization result just before surgery by the study coordinator.

Pre-operative examinations:

History summarizing previous surgical procedures, intraocular pressure while on treatment, target pressure at the discretion of the surgeon, visual field (SITA standard 24-2), gonioscopy, and a detailed description of the optic disc / nerve fiber layer by a glaucoma specialist was performed in all subjects included.

Post-operative examinations

Visits were undertaken at 1 day, 1 week, 2 weeks, 3 weeks, 1 month, 2 months, 3 months, 6 months, and 12 months.

Tests:

* visual fields (month 12)
* gonioscopy (month 12)
* intraocular pressure (all visits)
* optic disc examination (all visits, under dilation at 3 and 12 month)
* Pachymetry (preop exam)
* endothelial cell count (months 3 and 12)
* Bleb morphology (month 1 and 12)
* methodic registration of complications (all visits)

A specific CRF was designed with all variables and data required for the study which included a long list of individual potential complications

Pre-operative treatment. Prostaglandin analogues will be discontinued one week before surgery, but the rest of hypotensive drugs will be maintained until the day of surgery

Surgery. Each patient was assigned to one of the two arms (Ex-PRESS or Deep sclerectomy) the same day of surgery. The surgeon wil be informed of the randomization result just before surgery by the study coordinator.

The surgical technique is as follows: retro/peribulbar o subtenon's anesthesia, superior rectus or corneal traction suture, phacoemulsification through 2.1 to 2.8 mm incision with IOL implantation, a fornix-based conjunctival flap, sufficient but not excessive cauterization, application MMC 0,2 mg/ml for 2 minutes under the conjunctiva, then MMC was washed out with 50 ml of saline solution, then and according to the randomization result a scleral flap (5x5 mm in the NPDS, 4x4 mm in the Ex-Press group) is dissected.

Group 1. Then the Ex-PRESS device was placed according to the manufacturer's instructions and its position in the anterior chamber was verified by the surgeon.

Group 2. Deep sclerectomy (NPDS) was performed by dissecting a Deep scleral flap (4x4 mm) and peeling the trabeculo-descement membrane. A Esnoper (AJL, Vitoria, Spain) device was positioned under the external scleral flap and fixated with a 10/0 nylon suture.

Suture Nylon 10/00 suture was used to place four or five stitches in the Ex-Press group and 2 stitches in the NPDS group. Then a hermetic conjunctival suture was performed at the limbus with 10/0 nylon.

Post-operative treatment. All patients instilled Moxifloxacin Antibiotic every 6 hours for 1 week, Dexamethasone (every 2 hours for 1 month, every 4-6 hours on the second month and gradually tapered on the third month according to surgeon's instructions). Atropine was also used at the discretion of the surgeon when clinical finds recommended its use.

Suture lysis or gonio-punture were indicated and performed at the discretion of the surgeon, and they were always registered in the CRF.

Subconjunctival injections of anti-fibrotic agents and/or bleb needling were allowed and performed at the discretion of the surgeon.

DATA ANALYSIS Variables will be checked for normality using the Shapiro-Wilk test. The mean and standard deviation is going to be used to describe normally distributed variables which will be compared between independent groups using the Student t test. Variables that are found to be not normally distributed will be described by median and quartiles, and their comparison between independent groups wil be performed using the Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of open-angle glaucoma. Points a, b and c will be required:

   1. Glaucomatous visual field. Defined as the field presenting at least:

      * A group of 3 or more points with p < 5% in the pattern deviation map AND
      * One of them with a p < 1% in the pattern deviation map AND
      * Repeated in at least 2 VF.
   2. Glaucomatous optic nerve. Defined as the optic nerve observed in color photographs presenting:

      * Thinning of the neuroretinal rim that can be demonstrated by an alteration in the ISNT rule.
      * Presence of a notch "or"
      * Presence of papillary splinter hemorrhage "or"
      * Presence of a nerve fiber layer defect "or"
      * Cup to disc (C/D) ratio asymmetry > 0.3 that cannot be explained by asymmetry in the optic disc size "or"
      * C/D ratio > 0.8 that cannot be explained by a large optic disc size
   3. III or IV angle in Shaffer classification
2. Disease poorly controlled with medical treatment and/or laser at the discretion of the ophthalmologist (progression, higher than targeted pressure, poor compliance…)
3. Cataract with visual acuity between 0,1 (20/200) and 0.8 (20/25)

Exclusion Criteria:

1. Inflammatory, neovasular, closed-angle, normotensive glaucoma secondary to corticoids, or any type of glaucoma with advanced degree of functional lesion (Mean Defect < -20 dB)
2. Previous glaucoma surgery
3. Previous intraocular ocular surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-02; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | Up to 12 months
  mmHg

SECONDARY OUTCOMES:
Success rate at IOP <18 | Up to 12 months
  percentage of patients with < of 18 mmHg in intraocular pressure
Number of participants with adverse events assesed by questionare in case report file. | Up to 12 months
  Bullet list of complications to check for at each study visit from the date of randomization upt to 12 months
  List of complications in Case report file:
  Avascular bleb Bleb fibrosis Choroidal effusion Corectopia Corneal edema Corneal erosion Cystoid macular edema Descemet folds Epiretinal membrane Fibrin IOL Foreign body sensation Hematic tyndall Hypotony > 1 month Hypotony Maculopathy Iris incarceration Iris synechiae Lamellar macular hole Posterior capsule opacity Postoperative shunt closure Postoperative uveitis Seidel (early) Shallow anterior chamber Subconjunctival hemorrhage Tenon Cist Transient hypotony VA declined > 2 Snellen lines Vitreous in anterior chamber
Number of hypotensive medications needed | Up to 12 months
  Number of drugs prescribed by investigator to keep IOP under target from the date of randomization up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Antón, MD, PhD, Principal Investigator — Institut Catala de Retina
Locations (1):
- Institut Catala de Retina, Barcelona, Spain